CLINICAL TRIAL: NCT04992104
Title: Elucidating the Dynamics and Impact of the Gut Microbiome on Maternal Nutritional Status During Pregnancy
Brief Title: Microbiome and Malnutrition in Pregnancy
Acronym: MMIP
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Unity Health Toronto (Other); University of Toronto (Other); University of Calgary (Other); Dalhousie University (Other); Aga Khan University (Other); University of Alberta (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, John Parkinson, Senior Scientist, The Hospital for Sick Children
Other Study IDs: CTOREB3512; MRT-168043 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2021-06-16; First posted 2021-08-05 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy Related; Pregnancy Loss; Pregnancy Complications; Pregnancy; Parasitic Disease; Microbial Colonization; Microbial Disease; Parasitic Disease; Metabolomics; Malnutrition; Malnutrition, Infant; Malnutrition Pregnancy; Breast Feeding
MeSH Terms: conditions — Pregnancy Complications; Parasitic Diseases; Communicable Diseases; Malnutrition; Infant Nutrition Disorders; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The following samples will be collected: blood samples, stool samples and rectal swabs.
  Participants will have the option to have their blood samples biobanked for future genetic testing (This would be a separate study application in the future).
  More information on sample analysis can be found in section 10 of the protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is being conducted to investigate how a mother's nutritional status and her gut microbiome during pregnancy contribute to the birth outcomes and health of her baby. The gut microbiome is the totality of microorganisms (e.g. bacteria, viruses, fungi) living in the gastrointestinal tract. This study will focus on pregnant women, 28 years and younger living in the Toronto and greater Toronto area. The focus is on younger women due to their vulnerability to undernutrition. Pregnant participants, and upon delivery, their newborns will be followed throughout pregnancy and for a year afterwards. Throughout this period, the investigators will collect stool samples, rectal swabs, blood samples, health assessments, nutritional and dietary assessments and birth/ labour details. The goal is to define the relationship between a mother's nutritional status and her microbiome dynamics during pregnancy and how they contribute to the birth outcomes and growth of her newborn. With the hypothesis that alterations of the microbiota in the maternal gut (dysbiosis) exacerbated by nutritional status or pathogen exposure during pregnancy, impacts weight gain because of impaired nutrient absorption, leading to corresponding negative birth outcomes.

DETAILED DESCRIPTION:
This project represents the first systematic investigation of the impact of the microbiome on nutritional status during pregnancy in young women and directly aligns with global health initiatives focused on this vulnerable cohort. The goal of the study is to define the relationships between host nutritional status and microbiome dynamics during pregnancy and how they contribute to birth outcomes. The gut microbiome has a profound influence on host nutritional status. Dysbiosis (loss of diversity/beneficial microbes and gain of pathobionts) has emerged as a major factor in the development of undernutrition. Despite the importance of nutrition during pregnancy, few studies have examined the role of the microbiome on maternal health and birth outcomes. Further, little is known concerning the influence of enteric eukaryotic microbes, such as parasites, on the bacterial microbiome and host nutrition.

At the core of this study are two complementary cohorts of young women that provide an exceptional opportunity to obtain longitudinal samples to monitor the dynamic relationships between microbiome community structure and function with gut health and host nutritional status. This registration is for the the Toronto cohort of the study, which will focus on refugee and young adult obstetric clinics in Toronto, a population of specific relevance to undernutrition. This cohort is expected to yield insights into the influence of eukaryotic microbes that are often viewed as asymptomatic. The target demographic of the study is young mothers, 28 years of age and younger, in the Toronto and Greater Toronto Area. The investigators have identified this younger demographic due to the lack of knowledge on the microbiome of young women, and their vulnerability to undernutrition. A second complementary cohort will be based in the Matiari district of Pakistan. This project will yield unprecedented insights into the relationships between prokaryotic and eukaryotic microbes in the gut and their associations with maternal health and birth outcomes.

The central hypothesis of the study is that alterations of the microbiota in the maternal gut (dysbiosis) exacerbated by nutritional status or pathogen exposure during pregnancy, impacts weight gain because of impaired nutrient absorption, leading to corresponding negative birth outcomes.

The study will be a prospective, longitudinal, observational study to investigate the impact and relationship between prokaryotic and eukaryotic microbes in the gut and their association with maternal health and birth outcomes among young women, 28 years of age and younger in the Toronto and Greater Toronto Area. The study will aim to recruit 400 women into two groups based on BMI at time of recruitment (Normal BMI will be defined as between 20 and 24.9 kg/m2 and Low BMI will be defined as less than 20 kg/m2). With a goal of having 200 participants within the normal BMI group and 200 participants within the low BMI group. Although this is the recruitment aim, in the event that the investigators are unable to recruit 200 women with a low BMI, more women will be recruited that fall within the normal BMI range. The study will follow women and their infants over the course of their pregnancy and for a year post-partum, collecting stool, rectal and blood samples, nutritional information, heath assessments, anthropometric measurements and empowerment metrics at different time points.

ELIGIBILITY:
Inclusion Criteria:

1. Consent provided
2. Participant is between 8-20 weeks post-conception
3. Female aged 28 years of age and younger
4. Confirmation of pregnancy
5. Intend to comply with study procedures and follow up

Exclusion Criteria:

1. Women who do not meet the enrolment age criteria
2. Women who are 20 + weeks post-conception
3. Women who have taken antibiotics within the past 3 months Note: it is common practice to give the mother penicillin in perinatal period if they are GBS positive; because this is standardized across the board it would not act as an exclusion factor.

Max Age: 28 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Biological sex: as the study's primary aim is to investigate pregnancy, participation will be restricted to participants who are biologically female. However, the study is inclusive with respect to gender, including both cis-gendered and trans-gendered participants (biological female-to-male).
Study Population: The study population will consist of pregnant women, 28 years of age and younger, living in the Toronto and Greater Toronto Area. The investigators focus on younger women, due to the lack of knowledge about their microbiome and their vulnerability to undernutrition
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To assess if alterations of the microbiota in the maternal gut (dysbiosis) are associated with changes in maternal gestational weight gain. | 8-20 weeks post-conception, 30-34 weeks post conception
  The primary endpoint will be the change in maternal gestational weight gain (GWG) during pregnancy, measured between the first (8-20 weeks post-conception) and second time point (30-34 weeks post conception).

SECONDARY OUTCOMES:
Anthropometrics: Maternal BMI | 8-20 weeks post-conception, 30-34 weeks post-conception, delivery, 3-months post-partum, 6 months post-partum and 12 months post-partum
  calculated using weight and height; BMI = kg/m2
Anthropometrics: Maternal middle upper arm circumference | 8-20 weeks post-conception, 30-34 weeks post-conception, 3-months post-partum,and 12 months post-partum
  Measured in cm
Anthropometrics: Maternal triceps skinfold thickness | 8-20 weeks post-conception, 30-34 weeks post-conception, 3-months post-partum, and 12 months post-partum
  Measured in cm
Anthropometrics: Maternal height | 8-20 weeks post conception, 30-34 weeks post conception, delivery, 3 months post-partum and 12 months post partum
  Measured in cm
Anthropometrics: Maternal weight | 8-20 weeks post conception, 30-34 weeks post conception, delivery, 3 months post-partum and 12 months post-partum
  Measured in kg
Maternal blood biomarkers | 8-20 weeks post-conception, 30-34 weeks post-conception, and 12 months post-partum
  Concentration of HB + MCV, ferritin, and CRP
Infant blood biomarkers | 12 months
  Concentration of HB + MCV, ferritin, and CRP
Infant sex | Determined at delivery
  Female or Male
Infant morbidity | 3 months, 6 months and 12 months
  Assessed through infant health assessment questionnaires
Maternal morbidity | 8-20 weeks post-conception, 30-34 weeks post-conception, 3 months post-partum, 6 months post-partum and 12 months post-partum
  Assessed through health assessment questionnaires
Infant growth: weight | within 24 hours of birth, 3 months, 6 months and 12 months
  Measured in kg
Infant growth: length | within 24 hours of birth, 3 months, 6 months and 12 months
  Measured in cm
Infant growth: head circumference | within 24 hours of birth, 3 months, 6 months and 12 months
  Measured in cm
Infant growth: mid upper arm circumference | within 24 hours of birth, 3 months, 6 months and 12 months
  Measured in cm
Infant growth: triceps skinfold thickness | within 24 hours of birth, 3 months, 6 months and 12 months
  Measured in cm
Infant Gestational age | 8-20 weeks post conception
  Will be documented at baseline visit.
Breast feeding: amount and initiation of complementary feeding | within 24 hours of birth, 3 months, 6 months and 12 months
  Based off of WHO 2010 Guidelines: Indicators for assessing infant and young child feeding practices (Part 2 Measurement)
Maternal age | Documented at 8-20 weeks post-conception
  24 years or younger
Reported maternal medication use | 8-20 weeks post-conception, 30-34 weeks post-conception, within 24 hours of delivery, 3-months post-partum, 6 months post-partum and 12 months post-partum
  [Questionnaire]
Reported Infant medication use | within 24 hours of birth, 3 months, 6 months and 12 months
  [Questionnaire]
Maternal dietary intake | 8-20 weeks post conception, 30-34 weeks post conception and 12 months post partum
  Assessed through ASA 24 HR Dietary Recall system, completed 2x each time point
Dietary diversity | 8-20 weeks post conception, 30-34 weeks post conception, 3 months post-partum and 12 months post partum
  Minimum Dietary Diversity Score for Women (MDD-W)
Household annual food insecurity | 3 months post-partum and 12 months post-partum
  Food insecurity will be assessed using the Household Food Insecurity Access Scale (HFIAS)
Self-efficacy | 3 months post-partum and 12 months post partum
  Self-efficacy will be measured using the Generalized Self-Efficacy scale, developed by Schwarzer and Jerusalem
Perceived decision making | 3 months post-partum and 12 months post partum
  Questions pertaining to perceived decision-making are from the Pakistan Demographic and Health Survey (PDHS)
Perceived social support | 3 months post-partum and 12 months post partum
  Perceived social support will be measured using the Multi-dimensional Scale of Perceived Social Support (MSPSS), developed by Zimet et al.
Maternal demographics | 8-20 weeks post-conception
  Questions pertaining to demographic data are adapted from the Pakistan Demographic and Health Survey (PDHS)
Food insecurity | 8-20 weeks post conception, 3 months post partum and 12 months post partum
  Questionnaire developed by Hager, E.R., et al., Development and validity of a 2-item screen to identify families at risk for food insecurity.
Perceived parental stress | 3 months post-partum and 12 months post partum
  Perceived parental stress will be measured using the Perceived Stress Scale (PSS-10)
Preterm birth | Within 24 hours of birth
  noted in labor and birth chart review
Stillbirth | Within 24 hours of birth
  noted in labor and birth chart review
Small for gestational age | Within 24 hours of birth
  noted in labor and birth chart review
Large for gestational age | Within 24 hours of birth
  noted in labor and birth chart review
Birth size: length | within 24 hours of birth
  Measured in cm
Birth size: head circumference | within 24 hours of birth
  Measured in cm
Birth size: weight | within 24 hours of birth
  Measured in kg
Birth defects | within 24 hours of birth
  Assessed within 24 hours of birth
Delivery assessment | within 24 hours of birth
  Assessed within 24 hours of birth
Infant dietary intake: NutricheQ Questionnaire | 12 months
  NutricheQ questionnaire: a tool designed for toddlers aged 1 to 3 years of age, with a focus on markers for inadequate or excessive intake and dietary imbalances
Maternal stool biomarkers: Calprotectin, Lipocalin and Claudin 15 | 8-20 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum
  Markers in the stool for intestinal mass, inflammation, and gut permeability and circulating lipopolysaccharide, among other markers
Infant Stool biomarkers: Calprotectin, Lipocalin and Claudin 15 | 3 months and 12 months
  Markers in the stool for intestinal mass, inflammation, and gut permeability and circulating lipopolysaccharide, among other markers
Maternal: incidence of pathobionts | 8-20 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum
  As identified through 16S, 18S and ITS rDNA surveys
Infant: incidence of pathobionts | 3 months and 12 months
  As identified through 16S, 18S and ITS rDNA surveys
Maternal: metabolomic profile of stool (metabolites involved in central metabolism as analysed by Mass Spectrometry) | 8-20 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum
  Analysis of the core metabolites involved in central metabolism. These metabolites will be analysed through Mass Spec and include short chain fatty acids, amino acids, intermediates in energy metabolism and nucleotide biosynthesis
Maternal gut bacteria profile as measured through 16S rDNA sequence surveys | 8-20 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum
  measured through 16S rDNA sequence surveys
Maternal: blood metallomics profile as measured through ICP-MS (https://www.metabolomicscentre.ca/new_service/25) | 8-20 weeks post conception, 30-34 weeks post conception, and 12 months post partum
  TMIC Metallomics Platform to be used.
Infant: blood metallomics profile as measured through ICP-MS (https://www.metabolomicscentre.ca/new_service/25) | 12 months
  Through TMIC platform
Infant: gut bacterial profile as measured through 16S rDNA sequence surveys | 3 and 12 months post partum
  measured through 16S rDNA sequence surveys
Maternal metabolic pathway expression profile as measured through whole microbiome RNASeq (metatranscriptomics) | 8-20 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum
  measured through whole microbiome RNASeq (metatranscriptomics)
Infant eukaryotic microbiome profile as measured through 18S and ITS rDNA sequence surveys | 3 months and 12 months
  measured through 18S and ITS rDNA sequence surveys
Maternal eukaryotic microbiome profile as measured through 18S and ITS rDNA sequence surveys | 8-20 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum
  measured through 18S and ITS rDNA sequence surveys
Maternal bacterial gene expression profile as measured through whole microbiome RNASeq (metatranscriptomics) | 8-20 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum
  The output of these analyses are readouts of microbial gene expression detailing biochemical activities as well as the taxa responsible.
Maternal: microbiome taxonomic alpha and beta diversity | 8-20 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum
  To define taxonomic diversity, species profiles from 16S, 18S and ITS rDNA data will be clustered to identify differences in community structure across samples. Alpha diversity will be measured through indices such as Chao, Shannon and Simpson indices. Beta diversity will be measured through standard indices such as Bray-Curtis distances.
Infant: microbiome taxonomic alpha and beta diversity | 3 months and 12 months
  To define taxonomic diversity, species profiles from 16S, 18S and ITS rDNA data will be clustered to identify differences in community structure across samples. Alpha diversity will be measured through indices such as Chao, Shannon and Simpson indices. Beta diversity will be measured through standard indices such as Bray-Curtis distances.

CONTACTS AND LOCATIONS:
Overall Officials: John Parkinson, PHD, Principal Investigator — The Hospital for Sick Children; Shazeen Suleman, MD, Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - St. Michael's Hospital, Toronto
  - The Hospital for Sick Children, Toronto

IPD SHARING:
Plan to Share IPD: Yes
In addition to publishing findings in open access journals, the investigators will ensure all sequences and metabolomics datasets are deposited in appropriate public repositories. SOPs, pathogen samples and statistical methods developed through this project will be shared with the IMPACTT research core (https://www.impactt-microbiome.ca/). Microbiome sequence data will be uploaded on the National Centre for Biotechnology Information (NCBI).
  The NCBI acts as a central data repository for sequence data. In line with publication standards, the investigators are required to provide access to users who may wish to follow up on analyzing the microbiome data for their own purposes.
  The sample analysis information, including the sequencing data and metabolomics data will be de-identified and the patient sequence data will be removed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All sequence and metabolomics data will be made available within 12 months of study completion Supporting information will be shared at time of request
Access Criteria: Supporting information will be shared upon request Sequence and metabolomics datasets will be made available without restriction

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT04992104/Prot_SAP_002.pdf
  • Informed Consent Form (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT04992104/ICF_003.pdf